CLINICAL TRIAL: NCT05304520
Title: SISTER - Subcutaneous: Non-Interventional Study for Tysabri Patient Preference - Experience From Real World
Brief Title: A Study for Tysabri Participant Preference
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: DE-TYS-11923
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Relapsing-Remitting Multiple Sclerosis (RRMS)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- On Natalizumab: Switcher IV to SC Cohort: Participants who are already on natalizumab treatment, 300 milligrams (mg) IV infusion and who decide to switch to 2x150 mg SC injection administered as standard of care/routine clinical practice will be observed for up to 12 months.
  Interventions: Drug: Natalizumab
- Natalizumab-Naive IV Cohort: Participants who initiate natalizumab, 300 mg, IV infusion injection administered as standard of care/routine clinical practice will be observed for up to 12 months
  Interventions: Drug: Natalizumab
- Natalizumab-Naive SC Cohort: Participants who initiate natalizumab, 2x150 mg, SC injection administered as standard of care/routine clinical practice will be observed for up to 12 months.
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab — Administered as specified in the treatment arm.

SUMMARY:
The primary objective of this study is to collect, evaluate and compare data on participant preference between subcutaneous (SC) and intravenous (IV) natalizumab. The secondary objectives of this study are to evaluate the immunogenicity of SC natalizumab for natalizumab-naïve participants and collect and evaluate data on the multiple sclerosis (MS) disease-relevant parameters (relapse rate, time to first relapse, disability improvement and progression) over 12 months, in participants with natalizumab therapy starting on SC natalizumab or switching from IV natalizumab.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of highly active RRMS according to McDonald criteria (2018) and initiating natalizumab treatment is indicated based on current summary of product characteristics (SmPC)
* In RRMS participants who are already on natalizumab therapy, continued treatment must be indicated based on current SmPC

Key Exclusion Criteria:

* Progressive forms of MS
* Contraindication to natalizumab treatment according to natalizumab SmPC
* Concomitant treatment with other drugs for treating RRMS
* Participation in any interventional clinical trial NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with RRMS who are receiving or will initiate natalizumab (intravenous or subcutaneous) as standard of care/routine clinical practice will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants by Their Preferred Method of Natalizumab Administration at Month 6 | Month 6
  The participant preference will be measured by Patient preference questionnaire (PPQ) 1. PPQ 1 comprises of 3 questions - 1. "Are you satisfied with the route of administration of natalizumab?" (yes/no) and indicate main reason. 2. For SC participants only- "Have you experienced adverse events related to a subcutaneous injection." (1= mild to 5 = severe), and 3. "If you had to choose between subcutaneous or intravenous route again, which route would you choose?".
Number of Participants by Their Preferred Method of Natalizumab Administration at Month 12 | Month 12
  The participant preference will be measured by Patient preference questionnaire (PPQ) 1. PPQ 1 comprises of 3 questions - 1. "Are you satisfied with the route of administration of natalizumab?" (yes/no) and indicate main reason. 2. For SC participants only- "Have you experienced adverse events related to a subcutaneous injection." (1= mild to 5 = severe), and 3. "If you had to choose between subcutaneous or intravenous route again, which route would you choose?".

SECONDARY OUTCOMES:
Number of Participants Positive for Anti-Natalizumab-Antibody | Baseline, Month 6 and 12
Percentage of Participants Persistently Positive for Anti-Natalizumab-Antibody | Baseline, Month 6 and 12
Annual Relapse Rate | Baseline, Months 3, 6, 9, and 12
  An MS relapse is defined as the onset of new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings. Annual relapse rate is calculated as the total number of relapses in each treatment group adjusted for the duration of study treatment in person-years.
Time to Relapse | Baseline, Months 3, 6, 9, and 12
  An MS relapse is defined as the onset of new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings.
Number of Participants With Disability Improvement and Progression who Switch to Subcutaneous Natalizumab | Baseline, Months 3, 6, 9, and 12
  Progression is defined as an increase of at least 1.5 points from a baseline Expanded Disability Status Scale (EDSS) score of 0, or at least 1.0 point from a baseline EDSS score >0 and ≤5.5 points, or at least 0.5 point from a baseline EDSS score ≥6.0. EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) is reported. Improvement is defined analogously, and all other cases are considered as stable disease.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (40):
- Germany (40):
  - Neurozentrum am Königsplatz Augsburg; Dres. Müller und Schmid, Augsburg
  - Praxis Dr. Schöll, Bad Homburg
  - Caritas Krankenhaus Bad Mergentheim, Bad Mergentheim
  - Neurologische Praxis Dr. med. Boris-Alexander Kallmann, Bamberg
  - Marianne-Strauß-Klinik Starnberg, Berg
  - Neurologie am Mexikoplatz, Berlin
  - Neurologie im Tempelhofer Hafen Berlin, Berlin
  - Neurologisches Facharztzentrum Dr. Masri & Kollegen, Berlin
  - NFZB Neurologisches Facharztzentrum Berlin, Berlin
  - Praxis für Neurologie/Dr. med. Martin Delf, Berlin
  - Katholisches Klinikum Bochum gGmbH, Bochum
  - Praxis Dres. Kausch/Lippert, Bogen
  - Neurologische Studiengesellschaft Bonn GbR, Bonn
  - MVZ Daun GmbH, Daun
  - Neurologie Dillingen, Dillingen
  - Gemeinschaftspraxis für Neurologie, Düsseldorf
  - Praxis Dr. Hartmann, Eltville
  - Neuro Centrum science GmbH, Erbach im Odenwald
  - Universitätsklinikum Erlangen, Neurolische Klinik, Erlangen
  - med.ring GmbH, Essen
  - NeuroDot GmbH, Grevenbroich
  - GP Dr. med. Wolfgang Klostermann/ Dr. med. Samir Al-Boutros, Hagen
  - Krankenhaus Martha-Maria Halle-Dölau; Klinik für Neurologie, Halle
  - Universitätsklinikum Jena, Hans-Berger-Klinik für Neurologie, Jena
  - Praxis Dr. Fischer, Lappersdorf
  - Neurokomm - Gesellschaft für Studien und Kommunikation, Mannheim
  - NPS Neurologisch Psychiatrische Studiengesellschaft, Mannheim
  - GP Neurologie am Preußenmuseum/ Martina Lorenz/ Dr. med. Birgit Erker, Minden
  - Landesklinkum Mistelbach-Gänserndorf, Abteilung Neurologie, Mistelbach
  - Hygieia Pharmakologisches Studienzentrum Chemnitz GmbH, Außenstelle Mittweida, Mittweida
  - Amperklinikum München Haar, München
  - CODAST, München
  - Neurologie Neu-Ulm, Neu-Ulm
  - Bergmann.Consult, Neuburg am Inn
  - Neurozentrum Prien, Prien am Chiemsee
  - EMSA, Singen
  - NeuroSinsheim, Sinsheim
  - Nervenfachärztliche GP, Ulm
  - Neuropraxis München Süd, Unterhaching
  - Praxis Dr. Krause, Wolfratshausen

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Gold R, Schmidt S, Deisenhammer F, Motte J, Richter N, Taipale K, Salmen HC, Bohland C, Schirduan K. Real-world evidence and patient preference for subcutaneous versus intravenous natalizumab in the treatment of relapsing-remitting multiple sclerosis - initial results from the observational SISTER study. Ther Adv Neurol Disord. 2024 Apr 13;17:17562864241241382. doi: 10.1177/17562864241241382. eCollection 2024. PMID 38616781